CLINICAL TRIAL: NCT06256809
Title: Qualitative and Quantitative Analysis of Finger and Palmer Dermatoglyphics Traits in Potentially Malignant and Malignant Lesions of the Oral Cavity for Genetic Predilection: A Case-Control Study
Brief Title: Analyzing Handprint Patterns to Predict Oral Cancer Risks: A Comparative Study
Acronym: QQA-FPD-PMML
Status: Not yet recruiting | Type: Observational
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, Assistant Professor, King Khalid University
Other Study IDs: RGP1/347/44; RGP1/347/44 (Other Grant/Funding Number: King Khalid University)
Record Dates: First submitted 2024-02-01; First posted 2024-02-13 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Lesion Risk Assessment Group: This group comprises individuals undergoing evaluation for dermatoglyphic patterns indicative of a predisposition to oral premalignant and malignant lesions. The group includes two sub-cohorts: one consisting of patients with diagnosed oral conditions like Oral Leukoplakia (OL), Oral Submucous Fibrosis (OSF), and Oral Squamous Cell Carcinoma (OSCC), and a control sub-cohort of individuals without these conditions. Dermatoglyphic analysis, including qualitative (whorls, loops, arches) and quantitative (Total Finger Ridge Count (TFRC), atd angles) parameters, will be conducted to assess potential predictive patterns and their correlation with oral lesion risks. No direct interventions are involved; the study focuses on observation and pattern analysis for potential early diagnosis and risk assessment.
- Healthy Control Group: This group consists of individuals with no history or diagnosis of oral premalignant or malignant lesions. They serve as a baseline comparison to the "Oral Lesion Risk Assessment Group". The dermatoglyphic patterns (whorls, loops, arches) and quantitative parameters (Total Finger Ridge Count (TFRC), atd angles) of this group are analyzed and compared with those of the patient group to identify distinctive patterns or traits associated with oral health conditions. This comparison aims to enhance the understanding of dermatoglyphic variations and their potential role in predicting oral health risks. No interventions are involved; the group is purely observational for comparative analysis

SUMMARY:
Aims: To evaluate the qualitative and quantitative parameters of finger and palmar dermatoglyphic patterns in patients with oral premalignant and malignant lesions OBJECTIVES: 1. To record and study the palmar and fingerprint patterns in patients with oral premalignant and malignant lesions 2. To assess the variations in patterns of dermatoglyphic features between cases and controls and to observe the significant result.

3. To evaluate which dermatoglyphic pattern is predominant among patients with premalignant and malignant lesions.

Materials and METHODS: Fingerprints and palm prints were studied in 160 patients, who were randomly divided into four groups: A. 40 patients with a history of areca nut /tobacco intake with the occurrence of the premalignant lesion (B) 40 patients with a history of areca nut /tobacco intake with the occurrence of Oral Squamous Cell Carcinoma. (C) As healthy controls, 40 patients with tobacco/areca nut chewing habits, without any evidence of oral lesions (D) 40 patients without any habit, and without any oral lesions. Dermatoglyphic patterns were recorded and analyzed in the four groups using the standard ink method.

DETAILED DESCRIPTION:
The skin is the protective layer covering the entire human body which acts as a barrier against various pathogens and also acts as a thermoregulatory organ. Skin is covered with hair follicles and sebaceous glands except in the palmar aspect of hands and the plantar aspect of soles. Both regions of the human body are devoid of hair and sebaceous glands but these parts have increased nerve supply due to the presence of more sensory receptors.

A unique ridge pattern is present on the palmar aspect of hands and the plantar aspect of soles called Epidermal Ridges (ER). These ridges are unique/different for every individual. Primarily these ridges help in gripping the surface. After conception, this pattern starts to develop from the 7th to 21st week of intra-gestation life. Creating a certain manner of sweat gland pore arrangement around the Papilla (Conical eminence) leads to the formation of epidermal ridges and is completed by 52 days of the gestation period.

Various factors influenced the development of these pattern formations which include genetic and environmental factors. Abnormal configuration of dermal patterns is influenced by both genetic and environmental factors causing disturbance during the intrauterine gestation period of the fetus. One classic example of abnormal dermal patterns is associated with Down syndrome where there will be an alteration in the Ridge pattern due to retardation affecting the growth of different parts of bodies and ER.

The study of this variation of ER and fingertips of palm and sole is known as "Dermatoglyphics".

In Greek, Derma means 'skin' and Glyphic means 'curved'. The initiation of Dermatoglyphic was done by Sir Frank Galton and he classified it into three patterns: Loops, arches, and whorls. Harold Clements conducted the first study on genetic abnormality with Dermatoglyphics patterns in Down syndromes. The Father of dermatoglyphics is Cummins. J. CA Mayer in 1788 concludes in his study on fingerprint analysis that dermatoglyphics pattern cannot be duplicated in two individuals. In 1858, Sir William Herschel (British Chief Administrator of Officer in West Bengal) was the first to use dermatoglyphics for personal identification which was used for criminology. Patterns of Dermatoglyphics can influence the genetic makeup of an individual which can act as a guide for genetic diseases such as Down syndrome, Klinefelter's syndrome, cancer, Alzheimer's, ovarian cancer, and schizophrenia.

Fingerprints are different in each individual; these are inherited and permanent to one particular individual and do not repeat or change among parents, or siblings, not even in the monozygotic twins. Unless in case of severe burns, cuts, and bruises due to this. The preliminary feature of these fingerprints, they can be used as evidence for the identification of a person in the forensic department and can be used as a tool in many genetic abnormality studies.

Oral Leukoplakia (OL) and oral submucous fibrosis (OSF) are more common premalignant lesions with high risk of malignant transformation rates of 0.6 to 20% and 1.5 to 15% respectively.

Both lesions are majorly caused due to tobacco usage in different forms and associated with various features affecting oral mucosa like ulceration, xerostomia, burning sensation, and alteration in collagen deposition. These pre-malignant lesions of the oral cavity commonly lead to the formation of Oral squamous cell carcinoma (OSCC) due to alterations in the function of genes.

Human genes regulate Cell signaling and tumor suppression which contributes to a decrease in cancer cell production. The two main factors which influence most diseases are genetic and epigenetic. Development of oral or head and neck squamous cell carcinoma (HNSCC) is influenced by both these factors. Population-based studies to determine the genetic or familial disposition to oral cancers are limited by coexisting risk factors like smoking and alcohol. It is also believed that certain individuals inherit the susceptibility of inability to metabolize carcinogens or procarcinogens and/or an impaired ability to repair DNA damage. Oncogenes are altered growth-promoting regulatory genes that govern the cells' signal transduction pathways, and mutation of these genes leads to either overproduction or increased function of the excitatory proteins. Several oncogenes have been implicated in oral carcinogenesis. Aberrant expression of the proto-oncogene epidermal growth factor receptor (EGFR/c-erb 1), members of the ras gene family, c-myc, int-2, hst-1, PRAD-1, and bcl-1 is believed to contribute towards cancer development. Hence the study of these genetic functions and the abnormality of genes has a potential role in diagnosing the malignancy earlier. However, this procedure required for the assessment of genes is expensive and complex. Therefore assessing dermatoglyphics traits can be a simple, cost-effective, non-invasive procedure along with clinical features for the early diagnosis of cancer, OSCC, and pre-malignant lesions.

This study is conducted with the following objectives and aims:

1. To record and study the palmar and fingerprint patterns in patients with oral premalignant and malignant lesions.
2. To assess the variations in patterns of dermatoglyphic features between cases and controls and to observe the significant result.
3. To evaluate which dermatoglyphic pattern is predominant among patients with premalignant and malignant lesions.
4. To assess the usefulness of this technique in acting as a predictor of oral squamous cell carcinoma; the efficacy of this technique as a non-invasive diagnostic tool in the identification of oral squamous cell carcinoma patients and also to identify persons at risk of oral squamous cell carcinoma.

This study is assessed based on the following parameters: 1. Qualitative parameters: a. Whorls b. Loops c. Arches 2. Quantitative parameters: a. Total finger ridge count (TFRC) b. angle of the palm: at angles

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with specific oral conditions such as Oral Leukoplakia, Oral Submucous Fibrosis, or Oral Squamous Cell Carcinoma.
* Individuals willing to participate in the study.

Exclusion Criteria:

* Individuals with systemic diseases that could affect dermatoglyphic patterns.
* Individuals who have undergone treatments that could alter palmar or plantar patterns.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population for this type of research typically consists of individuals diagnosed with oral premalignant conditions like Oral Leukoplakia or Oral Submucous Fibrosis, and those with malignant lesions such as Oral Squamous Cell Carcinoma. A control group of individuals without these conditions is also included for comparison. The study aims to analyze and compare the dermatoglyphic patterns (fingerprints and palm prints) of these groups to explore potential indicators or predictors of oral health conditions.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Dermatoglyphic Pattern Types in Oral Lesion Patients | 6-12 months
  This measure will assess and document the prevalence of whorls, loops, and arches separately in the patient group, allowing for a direct comparison with the control group.and quantitative parameters (Total Finger Ridge Count (TFRC), atd angles) in patients with diagnosed oral premalignant (OL, OSF) and malignant lesions (OSCC). The primary outcome will evaluate the prevalence and characteristics of these patterns in the patient group compared to the control group.
Quantitative Dermatoglyphic Parameters in Oral Lesion Patients | 6-12 months.
  This measure will document the average TFRC and atd angles for the patient group, facilitating a comparison with average values from the control group to identify significant differences.

SECONDARY OUTCOMES:
Correlation between Dermatoglyphic Patterns and Severity of Oral Lesions | 6-12 months
  Assessing the relationship between the intricacy or uniqueness of dermatoglyphic patterns and the severity or stage of oral lesions. This measure aims to determine if more complex or distinct patterns are associated with more advanced or aggressive forms of oral conditions.

IPD SHARING:
Plan to Share IPD: Yes
Demographic Information: Age, gender, ethnicity, etc., ensuring individual anonymity.
  Clinical Data: Specifics of oral conditions, diagnosis details, and treatment histories.
  Dermatoglyphic Patterns: Detailed fingerprint and palm print patterns. Outcome Measures: Primary, secondary, and other specified outcomes from the study.
Supporting Information: Study Protocol, SAP, ICF
URL: http://notspecific